CLINICAL TRIAL: NCT04363918
Title: The Use of Bioelectrical Stimulation in the Treatment of Erectile Dysfunction: a Randomized Controlled Trial
Brief Title: The Use of Bioelectrical Stimulation in the Treatment of Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Cristiane Carboni, Professor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3.076.079
Record Dates: First submitted 2020-04-21; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention (IG1) (Active Comparator)
  Interventions: Device: bioelectric stimulation
- intervention (MyoStim group) (Active Comparator)
  Interventions: Device: bioelectric stimulation
- control (CG) (Sham Comparator)
  Interventions: Device: bioelectric stimulation

INTERVENTIONS:
Device: bioelectric stimulation — bioelectric stimulation

SUMMARY:
Erectile dysfunction (ED), as defined by the International Consultation on Sexual Medicine, is the consistent and recurrent inability to acquire or sustain an erection of sufficient rigidity and duration to engage in satisfactory sexual intercourse. In the search for other approaches to treat ED the use of bioelectrical stimulation (BES) has been successfully introduced and applied in clinical studies. In the search for other approaches to treat ED the use of bioelectrical stimulation (BES) has been successfully introduced and applied in clinical studies.

DETAILED DESCRIPTION:
The investigators randomized 30 male patients, aged 40 to 75 years, with known ED (defined as a score of less than 22 on the IIEF-5), who had been in a stable relationship for more than 6 months and not taking any ED medication.

Participants were randomly assigned to three groups: intervention (IG1), intervention (MyoStim group) or control (CG). The IG1 received FES therapy (50 Hz/500 μs) for a total of 4 weeks, divided into two weekly sessions lasting 15 minutes each, with intensity set lower than the motor threshold that was assessed individually. The MyoStim group received a combination of low frequency BES and microcurrente for a total of 4 weeks, divided in two weekly sessions lasting 45 minutes each with intensity set lower than the motor threshold that was assessed individually which was delivered via two patch electrodes placed on the dorsum surface of the penis and connected to a desk top Mettler model 240 Bioelectric Stimulator, which was adjusted to reach each of the signals included in the protocol. In all three groups two self-adhesive electrodes measuring 3 cm each were used. One electrode was placed at the base of the penis, while the second was attached 2 cm below the first one. The control group was treated with placebo FES machine (the red light functioning but there was no power). Both groups attended sessions twice a week for a period of 4 weeks, for a total of 8 FES sessions. Erectile function was assessed by the validated International Index of Erectile Function (IIEF-5) and Erection Hardness Score (EHS) instruments. All of the questionnaires were applied before and immediately after the treatment. The instruments were completed by a blinded investigator, according to the protocol to which the patient had been randomized. Only the physiotherapist who applied the technique was aware of group allocation. Participants had no treatment costs.

The IG1 received actual stimulation for only the VEGF signal during the each treatment period, while the multi-signal MyoStim group received actual stimulation at precise frequencies for the five proteins which were changed every 5-15 minutes including.

All subjects completed all 8 treatments and the study questionnaires and metrics of ED before and at the end of the study. The study was unblinded when the last enrolled patient had completed their 4 weeks of treatment. The study included an opportunity for all patients randomized to the Control group to then receive the full four-week, 8 session treatment, for whichever of the two active treatment arms, VEGF alone or Myostim, was shown to be most effective. MyoStim treatment was clearly superior to the other treatment arms and all ten Control subjects elected to complete the full 4-week treatment with the MyoStim protocol in an open-label cross-over design. These ten subjects were then added to the original cohort assigned to MyoStim, for a total of 20 patients in the MyoStim arm. The statistical analysis was completed for the original treatment assignments with 10 subjects in each group and the total of 20 MyoStim subjects versus VEGF alone or Control.

ELIGIBILITY:
Inclusion Criteria:

* men with known ED (defined as a score of less than 22 on the IIEF-5)
* who had been in a stable relationship for more than 6 months
* not taking any ED medication.

Exclusion Criteria:

* neurogenic ED (due to spinal cord injury, Parkinson's disease, multiple sclerosis, prostatectomy)
* hypogonadism (total testosterone < 300 ng/ dl)
* decompensated diabetes mellitus (fasting blood glucose > 200 mg/dl and/or glycated hemoglobin > 8%)
* decompensated systemic arterial hypertension (SBP > 160 and/or DBP > 100)
* morbid obesity
* diagnosis of coronary heart disease and/or cerebrovascular disease
* inability to understand the study objectives/technique or to provide informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Erectile function | 8 weeks
  Erectile Function With International Index of Erectile Function-5 Questionnaire: The IIEF-5 questionnaire score determined the presence and severity of ED: absent (> 21), mild (17-21), mild / moderate (12-16), moderate (8-11) and severe (<8)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Fornari, PhD, Study Chair — Federal University of Health Science of Porto Alegre
Locations (1):
- Mundo do Assoalho Pélvico, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No